CLINICAL TRIAL: NCT01966250
Title: Electroacupuncture as a Complement to Usual Care for Patients With Non-acute Pain After Back Surgery: a Study Protocol for a Pilot Randomized Controlled Trial
Brief Title: Electroacupuncture as a Complement to Usual Care for Patients With Non-acute Pain After Back Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korean Medicine Hospital of Pusan National University (Other)
Responsible Party: Principal Investigator, Byung-Cheul Shin, associate professor, Korean Medicine Hospital of Pusan National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013012; K13273 (Other Grant/Funding Number: Korea Institute of Oriental Medicine)
Record Dates: First submitted 2013-10-11; First posted 2013-10-21 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Low Back Pain; Pain, Postoperative; Failed Back Surgery Syndrome
MeSH Terms: conditions — Low Back Pain; Pain, Postoperative; Failed Back Surgery Syndrome | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Electroacupuncture and Usual care (Experimental): 15 minutes of electroacupuncture and usual care. Usual care contains 15 minutes ICT(Interferential Current Therapy), 10 minutes hot pack or ice pack and education of patients.
  Interventions: Device: electroacupuncture and usual care
- usual care (Active Comparator): 15 minutes ICT, 10 minutes hot pack or ice pack and education of patients
  Interventions: Device: Usual care

INTERVENTIONS:
Device: electroacupuncture and usual care — Electroacupuncture: Using 0.25 mm (diameter) X 0.40 mm (length) sized disposable stainless steel needles, electric stimulation will be applied with an electronic stimulator (ES-160, ITO co. LTD, Japan) 2 times/week × 4 weeks. Stimulation will be applied with the current in biphasic wave form. Acupuncture points are Jia-ji (Ex-B2, L3-L5; bilateral) as necessary points and reasonable points (according to decision of practitioner) as accessory points. Each session lasts 15 minutes.
  Usual care: Physical therapy and patient education will be performed 2 times per week for 4 weeks. ICT lasts 15 minutes and Hot or Ice pack lasts 10minutes. Doctors will educate patient physiology, pathology, and epidemiology of low back pain. And also suitable postures and exercises for low back pain will be educated.
  Arms: Electroacupuncture and Usual care
Device: Usual care — Usual care: Physical therapy and patient education will be performed 2 times per week for 4 weeks. ICT lasts 15 minutes and Hot or Ice pack lasts 10minutes. Doctors will educate patient physiology, pathology, and epidemiology of low back pain. And also suitable postures and exercises for low back pain will be educated.
  Arms: usual care

SUMMARY:
The purpose of this study is to find out the effectiveness of integrative medicine model for pain relief and improvement of function and quality of life on the patients with pain after back surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose low back pain persisted or recurred after back surgery with or without leg pain.
* Patients whose pain has been persisted at least 3 weeks recently and who are necessary to care intermittent medical treatments (eg. medication, injection, physio therapy).
* Patients with pain, defined as an Visual Analogue Scale (VAS) value ≥ 50mm.
* Patients who are 19 - 70 years of age.
* Patients who agreed to voluntarily participate in this study and signed informed consent.

Exclusion Criteria:

* Patients who have been diagnosed with a serious disease that can cause low back pain (e.g., cancer, vertebral fracture, spinal infection, inflammatory spondylitis, cauda equine compression, or other disqualifying conditions).
* Patients with progressive neurological deficit or severe neurological symptoms.
* Patients whose pain causes are not resulted from spine or resulted from soft tissue diseases(e.g., cancer, fibromyalgia, rheumatoid arthritis, gout).
* Patients with a chronic disease that could influences the effects of the treatment or the analysis of treatment results (e.g., cardiovascular disease, diabetic neuropathy, fibromyalgia, rheumatoid arthritis, dementia, epilepsy, or other disqualifying conditions).
* Patients for whom acupuncture would be inappropriate or unsafe (e.g., hemorrhagic disease, clotting disorders, a history of receiving anticoagulant therapy, severe diabetes with a risk of infection, severe cardiovascular disease, or other disqualifying conditions)
* Patients who are currently pregnant or planning the pregnancy.
* Patients with psychiatric diseases.
* Patients who are participating in other clinical trial.
* Patients who are unable to sign informed consent.
* Patients who are judged to be inappropriate for the clinical study by the researchers, such as inability to read and write Korean.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | up to 4 months

SECONDARY OUTCOMES:
Oswestry Disability Index | up to 4 months
EuroQoL 5-Dimension Questionnaire | up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Byung-cheul Shin, Principal Investigator — Pusan National University Korean Medicine Hospital
Locations (1):
- Pusan National University Korean Medicine Hospital, Yangsan, Gyeongsangnam-do, South Korea

REFERENCES:
- [Derived] Heo I, Hwang MS, Hwang EH, Cho JH, Ha IH, Shin KM, Lee JH, Kim NK, Son DW, Shin BC. Electroacupuncture as a complement to usual care for patients with non-acute low back pain after back surgery: a pilot randomised controlled trial. BMJ Open. 2018 May 17;8(5):e018464. doi: 10.1136/bmjopen-2017-018464. PMID 29773696
- [Derived] Hwang MS, Heo KH, Cho HW, Shin BC, Lee HY, Heo I, Kim NK, Choi BK, Son DW, Hwang EH. Electroacupuncture as a complement to usual care for patients with non-acute pain after back surgery: a study protocol for a pilot randomised controlled trial. BMJ Open. 2015 Feb 4;5(2):e007031. doi: 10.1136/bmjopen-2014-007031. PMID 25652804